CLINICAL TRIAL: NCT01730560
Title: Rehabilitation For Acquired Visual Field Defects: Development Of A Bottom-Up Approach
Acronym: VISIOTRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2010.615; 2010-A00702-37 (Other: ID-RCB)
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Acquired Visual Field Defects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1:Treatment A (Experimental): Treatment A (active) followed by treatment B (neutral)
  Interventions: Other: Treatment A
- Arm 2: Treatment B (Experimental): Treatment B (neutral) followed by treatment A (active)
  Interventions: Other: Treatment B

INTERVENTIONS:
Other: Treatment A — The computer-based training task consists of a novel ramp-step search paradigm with a stimulus traversing the screen from left to right or right to left. Subjects are asked to pursue the stimulus (ramp phase) and then saccade to find its location when it suddenly jumps (step phase). The stimulus is an open spinning circle. At the end of each movement, the gap can be located at the top or at the bottom, and patients are asked to indicate this location by pushing the response button as quickly as possible.
  The starting point will alternate between left and right. The training task includes 3 sessions with 100 movements each. Reaction Times and errors will be monitored online to ensure that the patient performs the task correctly.
  Each treatment phase has the same pattern:
  * two visits in pre-tests evaluation (V1 and V2),
  * one visit to perform treatment (A or B) and to assess immediate and 2h post-effects (V3),
  * two visits after treatment (V4 at one week and V5 at one month).
  Arms: Arm 1:Treatment A
Other: Treatment B — Placebo treatment using the same computer-based training task, but including only the ramp phase.
  Each treatment phase has the same pattern:
  * two visits in pre-tests evaluation (V1 and V2),
  * one visit to perform treatment (A or B) and to assess immediate and 2h post-effects (V3),
  * two visits after treatment (V4 at one week and V5 at one month).
  Arms: Arm 2: Treatment B

SUMMARY:
Cortical Visual Field Defects (CFVD) are common after acquired brain injury. They often cause problems with reading and visual exploration which impact on patients' quality of life. Apart from the substitutive method that uses prisms directly placed on glasses, two main rehabilitative methods have been explored previously: one restorative and one compensatory. The most effective methods seem to be based on compensatory training paradigms that target eye movements. They rely on voluntary mass-practice that induces changes in exploratory saccadic behaviour, particularly into the blind hemifield. Previous studies using this method have shown changes in visual scanning patterns but with only a marginal profit in terms of functional benefit.

In the present study, the investigators developed a new approach to the compensatory visual field training based solely on a bottom-up mechanism. It does not require the patients' ability to voluntarily maintain attention oriented to the affected field, which may be difficult for brain-damaged patients. As previously reported in other pathological contexts (e.g. use of prism adaptation or sensory stimulation in neglect patients), bypassing voluntary and conscious implication of the patient can produce improvements by a more automatic process.

The investigators hypotheses are: 1) that a novel ramp-step search paradigm can be used by hemianopic patients to automatically improve targeted eye movements into their blind visual field; and 2) that this will lead to behavioural improvements on ecologically valid tests of visual search.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female
* Stroke (ischemia or hemorrhage) documented by CTscan or MRI
* Traumatic brain injury (TBI) documented by CTscan or MRI
* Right or Left hemianopia defined by perimetry
* All subjects must be between the ages of 18-80
* Aetiology of visual field defect : Stroke (ischemia or hemorrhage)
* Delay post-stroke : at least 6 months
* Only one lesion on CTscan or MRI (performed in a maximal delay of 6 months)
* Corrected monocular visual acuity > 5/10
* Possible understanding of experimental conditions
* Patient being able to be quiet and sit during at least 2 hours
* Having given written informed consent prior to any procedure related to the study
* Availability for the period of the study
* Covered by a Health System where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research

Exclusion Criteria:

* Ophthalmologic criteria : monocular visual acuity < 4/10, strabismus , diplopia , ocular instability , nystagmus, maculopathy , glaucoma , retinopathy , orthoptic rehabilitation
* Neurologic criteria : sever phasic disturbances , neurologic degenerative affection , non controlled seizure , severe handicap non compatible with prolonged sit position or concentration during 30 consecutive minutes
* No command of french language
* Non stabilized medical situation
* Females who are pregnant, nursing, or planning a pregnancy during the study period, or females of childbearing potential, not using a reliable means of contraception.
* Not under any administrative or legal supervision

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-11-29 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2018-06-13 (Actual)

PRIMARY OUTCOMES:
Difference in performance (mean reaction time - RT) of an ecological visual search task between pre-tests and immediate post-test for each patient according to treatment (A or B). | 1 week

SECONDARY OUTCOMES:
Errors and omissions at each evaluation session for the visual search task | 1, 2 and 5 weeks
  Mean RT difference, errors and omissions at several visual tasks (rapid scanning task, exploratory visual tasks, reading task) at each evaluation session Parameters of visual field perimetry before and after treatment Oculo-motor parameters during the different tasks (i.e. amplitude and latencies for saccades and fixations)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Jacquin-Courtois, MD, PhD, Principal Investigator — Service de Médecine Physique et de Réadaptation
Locations (1):
- Service de Médecine Physique et de Réadaptation,Hôpital Henry Gabrielle, Saint-Genis-Laval, France

REFERENCES:
- [Background] Ong YH, Jacquin-Courtois S, Gorgoraptis N, Bays PM, Husain M, Leff AP. Eye-Search: A web-based therapy that improves visual search in hemianopia. Ann Clin Transl Neurol. 2015 Jan;2(1):74-8. doi: 10.1002/acn3.154. Epub 2014 Nov 27. PMID 25642437